CLINICAL TRIAL: NCT01499953
Title: Superficial Vein Thrombosis (SVT) Treated for Forty-five Days With Rivaroxaban Versus Fondaparinux
Brief Title: Superficial Vein Thrombosis (SVT) Treated With Rivaroxaban Versus Fondaparinux
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GWT-TUD GmbH (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SURPRISE-2011
Record Dates: First submitted 2011-12-19; First posted 2011-12-26 (Estimated); Results first posted 2023-05-15 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2022-07

CONDITIONS: Superficial Vein Thrombosis
Keywords: superficial vein thrombosis; thrombosis; SVT
MeSH Terms: conditions — Thrombosis | interventions — Rivaroxaban; Fondaparinux

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rivaroxaban (Experimental): Rivaroxaban for 45 days oral dose: 10 mg OD
  Interventions: Drug: Rivaroxaban
- Fondaparinux (Active Comparator): Fondaparinux for 45 days subcutaneous application: 2,5 mg OD
  Interventions: Drug: Fondaparinux

INTERVENTIONS:
Drug: Rivaroxaban — Dose: 10 mg Duration: 45 (±5) days Frequency: once daily Application: oral
  Other Names: Xarelto
  Arms: Rivaroxaban
Drug: Fondaparinux — Fondaparinux Dose: 2.5 mg Duration: 45 (±5) days Frequency: once daily Application: subcutaneous
  Other Names: Arixtra
  Arms: Fondaparinux

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of rivaroxaban versus fondaparinux in the treatment of superficial vein thrombosis (SVT).

DETAILED DESCRIPTION:
Evaluation of efficacy and safety of 45 days of rivaroxaban 10 mg vs. fondaparinux 2.5 mg in the treatment of superficial vein thrombosis of risk patients for major VTE complications to prove non-inferiority of oral rivaroxaban treatment

ELIGIBILITY:
Inclusion Criteria:

* acute symptomatic supragenual superficial vein thrombosis of the leg
* at least one of the following major risk factor for VTE:
* age > 65 years or
* male sex or
* history of DVT/PE/SVT or
* history of cancer or active cancer or
* autoimmune disease or
* SVT of a non-varicose vein
* thrombus extension of at least 5 cm
* proximal thrombus end with more than 3 cm distance to the saphenofemoral junction (SFJ)
* age > 18 years
* written informed consent

Exclusion Criteria:

* other indication for therapeutic anticoagulation such as acute deep vein thrombosis, acute pulmonary embolism, atrial fibrillation with indication for anticoagulant therapy
* any PE or DVT within last 6 months before inclusion
* clinical signs of PE without objective exclusion (CT or VQ scan, angiography)
* SVT without signs of thrombotic/inflammatory activity (activity signs: diameter > 4 mm, pain, redness, elevated local or systemic temperature)
* SVT after sclerotherapy
* Duration of symptoms > 3 weeks
* pretreatment of more than 72 h with therapeutic dosages of oral or parenteral anticoagulants
* pretreatment of more than 5 days with subtherapeutic oral or parenteral anticoagulants
* indication for escalated antiplatelet therapy (monotherapy with aspirin > 325 g/d and any dual antiplatelet therapy)
* SVT closer than 3 cm to saphenofemoral junction (SVJ)
* anticipated superficial vein surgery within 90 days
* anticipated thrombolytic therapy within 90 days
* manifest clinically relevant bleeding
* clinically relevant bleeding in the last 30 days before study inclusion
* major surgery within last 30 days before inclusion
* ophthalmic, spinal or cerebral surgery within last 90 days
* severe head trauma within last 90 days
* hemorrhagic stroke within last 12 months
* hereditary or acquired severe hemorrhagic diathesis
* gastrointestinal bleeding within last 90 days requiring endoscopy
* uncontrolled arterial hypertension (systolic > 180 mm Hg, diastolic > 110 mm Hg)
* acute endocarditis
* low platelet count (< 100 x 109/l)
* Prothrombin time < 50 %
* calculated creatinine clearance < 30 ml/min
* significant liver disease such as acute hepatitis, chronic active hepatitis, cirrhosis
* life expectancy < 3 months
* any contraindications listed for rivaroxaban or fondaparinux
* women of child bearing potential without safe contraception method
* pregnant or breastfeeding women
* participation in another trial with pharmacological intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 472 (Actual)
Dates: Start 2012-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Beyer-Westendorf, MD, Principal Investigator — on behalf of GWT-TUD GmbH
Locations (23):
- Germany (23):
  - Hautarztpraxis, Freiburg im Breisgau, Baden-Wurttemberg
  - Gemeinschaftspraxis Mietaschk, Bilderling, Kaiser, Tato, München, Bavaria
  - Chriurgische Praxisklinik, Baesweiler, North Rhine-Westphalia
  - Krankenhaus Dresden-Friedrichstadt, Dresden, Saxony
  - Universitätsklinikum Dresden, Dresden, Saxony
  - Oberlausitz-Gefäßpraxis, Görlitz, Saxony
  - Franziskus-Krankenhaus Berlin, Berlin
  - MVZ Ramdohr, Praxis für Cardiovaskulär- u. Ultraschalldiagnostik, Berlin
  - Praxis für Chirurgie & Gefäßmedizin, Berlin
  - Praxis für Allgemeinmedizin und Phlebologie, Cologne
  - Klinikum Darmstadt GmbH, Darmstadt
  - Gemeinschaftspraxis Eggeling und Winter, Eschwege
  - Asklepios Westklinikum Hamburg, Hamburg
  - Universitätsklinikum Heidelberg, Heidelberg
  - Internistische Praxisgemeinschaft, Hoppegarten
  - Akademie für Gefäßkrankheiten e.V., Karlsbach
  - Universitätsklinikum Leipzig AöR Innere Medizin - Angiologische Ambulanz, Leipzig
  - Universitätsklinikum Schleswig-Holstein, Campus Lübeck, Lübeck
  - Praxis Dr. Franke, Magdeburg
  - Kardiologie Mühldorf am Inn, Mühldorf
  - Praxis Dr. Kähler, Rostock
  - Praxis für Gefäßmedizin am Tegernsee, Rottach-Egern
  - Venenzentrum Wiesbaden, Wiesbaden

REFERENCES:
- [Derived] Kearon C, Carrier M, Gu CS, Schulman S, Bates SM, Kahn SR, Chagnon I, Nguyen DT, Wu C, Rudd-Scott L, Julian JA. Rivaroxaban Compared to Placebo for the Treatment of Leg Superficial Vein Thrombosis: A Randomized Trial. Semin Thromb Hemost. 2020 Nov;46(8):977-985. doi: 10.1055/s-0040-1718891. Epub 2020 Dec 23. PMID 33368114
- [Derived] Beyer-Westendorf J, Schellong SM, Gerlach H, Rabe E, Weitz JI, Jersemann K, Sahin K, Bauersachs R; SURPRISE investigators. Prevention of thromboembolic complications in patients with superficial-vein thrombosis given rivaroxaban or fondaparinux: the open-label, randomised, non-inferiority SURPRISE phase 3b trial. Lancet Haematol. 2017 Mar;4(3):e105-e113. doi: 10.1016/S2352-3026(17)30014-5. Epub 2017 Feb 16. PMID 28219692
- [Derived] Werth S, Bauersachs R, Gerlach H, Rabe E, Schellong S, Beyer-Westendorf J. Superficial vein thrombosis treated for 45 days with rivaroxaban versus fondaparinux: rationale and design of the SURPRISE trial. J Thromb Thrombolysis. 2016 Aug;42(2):197-204. doi: 10.1007/s11239-016-1354-3. PMID 26973347

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 25th April 2012 through 18th February 2016, a total of 485 patients were screened at 23 study sites in Germany. Of them, 9 patients did not meet the eligibility criteria. For another 4 subjects, signatures either on informed consent form or data protection waiver were not provided and therefore, these 4 subjects were not included in the study.
Pre-assignment Details: 472 patients were randomized to one of the two treatment groups. One patient in the fondaparinux group withdrew consent after randomization but before the first study drug administration.
Period: Overall Study
Arm/Group | Fondaparinux | Rivaroxaban
Started | 236 | 236
Participants Who Received at Least One Dose of Study Medication | 235 | 236
Completed | 226 | 222
Not Completed | 10 | 14

BASELINE CHARACTERISTICS:
Population: Safety analysis set (Per protocol analysis set for risk factors)
Groups:
- Total: Total of all reporting groups
Arm/Group | Rivaroxaban | Fondaparinux | Total
Number analyzed (Participants) | 236 | 235 | 471
Age, Continuous [Mean (Full Range); unit: years] | 60.7 [21 to 94] | 59.8 [23 to 92] | 60.3 [21 to 94]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136 | 148 | 284
  Male | 100 | 87 | 187
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian | 233 | 234 | 467
  Race: Other | 3 | 1 | 4
Weight [Mean (Full Range); unit: kg] | 86.2 [50 to 145] | 88.0 [50 to 165] | 87.1 [50 to 165]
Height [Mean (Full Range); unit: cm] | 170 [147 to 196] | 171 [150 to 200] | 170 [147 to 200]
BMI [Mean (Full Range); unit: kg/m^2] | 29.8 [18.7 to 53.8] | 30.2 [17.7 to 64.9] | 30.0 [17.7 to 64.9]
Risk factors [Count of Participants; unit: Participants] — Population: Number of patients with specific risk factors was evaluated for the per protocol analysis set only.
  Participants
    Age > 65 years: number analyzed (Participants) | 211 | 224 | 435
    Age > 65 years | 82 | 84 | 166
    History of cancer or active cancer: number analyzed (Participants) | 211 | 224 | 435
    History of cancer or active cancer | 16 | 21 | 37
    Autoimmune disease: number analyzed (Participants) | 211 | 224 | 435
    Autoimmune disease | 3 | 4 | 7
    SVT of non-varicose vein: number analyzed (Participants) | 211 | 224 | 435
    SVT of non-varicose vein | 60 | 72 | 132
    Male: number analyzed (Participants) | 211 | 224 | 435
    Male | 89 | 84 | 173
    History of DVT/PE/SVT: number analyzed (Participants) | 211 | 224 | 435
    History of DVT/PE/SVT | 105 | 106 | 211

OUTCOME MEASURES:

1. Primary Outcome: Rate of Objectively Confirmed VTE Complications
Description: The primary efficacy outcome was the composite of death from any cause, symptomatic pulmonary embolism (confirmed by ventilation-perfusion scanning, helical computed tomography, pulmonary angiography, or autopsy), symptomatic deep vein thrombosis (confirmed by ultrasonography or venography), or symptomatic extension towards the saphenofemoral junction or symptomatic recurrence of superficial vein thrombosis (confirmed by ultrasonography) up to day 45.
Time Frame: 45 +/- 5 days
Population: Per protocol set
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban | Fondaparinux
Number analyzed (Participants) | 211 | 224
Participants | 7 | 4
Statistical Analysis 1: Comparison: Rivaroxaban vs Fondaparinux; Test type: Non-Inferiority — The hypotheses for non-inferiority test using ∆=4.5% for the difference between incidence rates were H0: πrivaroxaban-πfondaparinux ≥ 4.5%, H1: πrivaroxaban-πfondaparinux < 4.5% where πfondaparinux and πrivaroxaban were the incidence rates of CIAC confirmed VTE complications up to Day 45 in the treatment groups. Rejection of the null hypothesis would have concluded that rivaroxaban was not inferior to fondaparinux. To calculate the p-value, an asymptotic test for non-inferiority was used; p = 0.0252, asymptotic test for non-inferiority

2. Secondary Outcome: Composite Primary Efficacy Outcome
Description: For this, secondary efficacy outcomes were the composite primary efficacy outcome up to Day 90 and the following outcomes up to Day 45 and Day 90: each component of the primary efficacy outcome, the rate of major VTE (composite of symptomatic pulmonary embolism or symptomatic proximal DVT or VTE-related death) and the rates of surgery for SVT.
Time Frame: 90 +/- 10 days
Population: Per protocol analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban | Fondaparinux
Number analyzed (Participants) | 211 | 224
Participants | 15 | 15

3. Secondary Outcome: Rate of Major VTE
Description: composite of:
  * symptomatic pulmonary embolism
  * symptomatic proximal DVT
  * VTE-related death
Time Frame: 90 +/-10 days
Population: Per protocol set
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban | Fondaparinux
Number analyzed (Participants) | 211 | 224
Participants
  Deep vein thrombosis | 6 | 2
  Pulmonary embolism | 0 | 0
  VTE-related death | 0 | 0

4. Secondary Outcome: Rates of Surgery for SVT
Time Frame: 90 +/-10 days
Population: Per protocol set
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban | Fondaparinux
Number analyzed (Participants) | 211 | 224
Participants | 0 | 2

5. Other Pre Specified Outcome: Major Bleeding (Main Safety Outcome)
Description: * associated with a fall of hemoglobin of 2 g/l or more, or;
  * leading to a transfusion of 2 or more units of packed red blood cells or whole blood, or;
  * occurring into a critical site such as intracranial, intraspinal, intraocular, pericardial, intraarticular, intramuscular with compartment syndrome, retroperitoneal, or;
  * fatal bleeding.
Time Frame: 45 +/- 5 days
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban | Fondaparinux
Number analyzed (Participants) | 236 | 235
Participants | 0 | 0

6. Other Pre Specified Outcome: Clinically Relevant Non-major, Minor and Total (Any) Bleeding
Description: Clinically relevant, non-major bleeding is defined as any overt bleeding and
  * associated with a medical intervention, or
  * unscheduled contact with the physician (presence or telephone contact)
  * temporary or complete cessation of study drug
  * associated with any relevant discomfort to the patient (pain, impairment of activities of daily life)
Time Frame: 45 +/- 5 days
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban | Fondaparinux
Number analyzed (Participants) | 236 | 235
Participants
  CRNM bleeding | 6 | 1
  Minor bleeding | 15 | 15
  Any bleeding | 20 | 16

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are reported between first study drug administration until 5 days after last study drug administration.
Arm/Group | Fondaparinux | Rivaroxaban
All-Cause Mortality (participants affected / at risk) | 0/235 | 1/236
Serious Adverse Events (participants affected / at risk) | 3/235 | 7/236
Other Adverse Events (participants affected / at risk) | 0/235 | 0/236
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fondaparinux (N=235) | Rivaroxaban (N=236)
Suspected infection-associated seizure (Infections and infestations) | 0 (0) | 1 (1)
Lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Mucosal bleeding (General disorders) | 0 (0) | 1 (1)
New onset of atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Worsening of arterial hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hemorrhagic allergic skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Diabetic foot syndrome with tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Hospitalisation for COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Transient ischemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Sigmoid diverticulitis (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes